CLINICAL TRIAL: NCT03912753
Title: Building Mobile HIV Prevention and Mental Health Support in Low-resource Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Yale University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Corina Lelutiu-Weinberger, Associate Professor of Health Sciences Research (in Nursing), Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAU2518; R01MH116829 (NIH)
Record Dates: First submitted 2019-04-02; First posted 2019-04-11 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Human Immunodeficiency Virus; Risk Reduction; Alcohol Abuse; Depression, Anxiety; Behavior, Sex
Keywords: HIV; Syphilis; Chlamydia; Gonorrhea
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Risk Reduction Behavior; Alcoholism; Depression; Anxiety Disorders; Sexual Behavior; Syphilis; Chlamydia Infections; Gonorrhea

STUDY DESIGN:
Intervention Model Description: The investigators will recruit, screen, assess, and randomize gay and bisexual men at risk for HIV infection and alcohol abuse to either the Comunică intervention (n=163) or EAC (n=163).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comunică (Experimental): Comunică is delivered over eight 60-min live chat sessions, delivered by trained psychologists, on our mHealth study platform compatible with any mobile device (laptops, smartphones).
  Interventions: Behavioral: Comunică
- Education Attention Control (EAC) (Active Comparator): The EAC condition consists of eight self-administered modularized topics, content-matched with the Comunică sessions, which we have generated based on our HIV-prevention education with GBM in the US and Romania.Topics include 1) GBM identity, 2) "HIV 101," 3) HIV/STI testing, 4) alcohol and the body, 5) the role of alcohol in HIV risk, 6) HIV-status disclosure and sexual health communication, 7) finding social supports, and 8) summary. EAC participants will receive five quiz questions after each module, with correct answers in a following screen.
  Interventions: Other: Education Attention Control

INTERVENTIONS:
Behavioral: Comunică — Comunică is based on the Information-Motivation-Behavioral Skills (IMB) model of health behavior change, which postulates that individuals must possess the requisite information for enacting sexual health, motivation to change their HIV risk and alcohol use, and behavioral skills necessary for reducing their risk. Therefore, Comunică includes MI to provide accurate information about HIV transmission, alcohol abuse, and local GBM-affirmative health resources and build motivation to improve behavioral skills (via CBST). CBST is a therapeutic approach used in the treatment of various behavioral problems, such as alcohol abuse and depression and more recently HIV risk. CBST can help modify cognitions driving unhealthy behaviors, promote awareness of contextual triggers and unhealthy behavioral patterns, and teach coping skills to improve health. Comunică also draws upon minority stress theory recognizing that stigmatizing societal contexts compromise health behavior.
  Arms: Comunică
Other: Education Attention Control — The EAC condition consists of eight self-administered modularized topics, content-matched with the Comunică sessions, which we have generated based on our HIV-prevention education with GBM in the US and Romania.
  Arms: Education Attention Control (EAC)

SUMMARY:
The purpose of this research study is to provide help and support for mental health and human immunodeficiency virus (HIV) risk reduction among Romanian gay and bisexual men.

GBM will participate in this study using mobile device (phones, tablets, or laptops) and will complete several confidential surveys and 8 confidential one-hour sessions, either with a trained counselor via chat or by reading about health information. This study also involves testing for HIV, syphilis, chlamydia, and gonorrhea.

DETAILED DESCRIPTION:
This project is designed to remedy unaddressed and interlocking HIV-prevention and mental health needs among gay and bisexual men (GBM) in the Central Eastern European country of Romania, and their underpinning stigma-related mechanisms. Rampant stigma contributes to the increasing prevalence of HIV among Romanian GBM (from under 10% in 2009 to close to 20% in 2014, by best available estimates) and keeps GBM out-of-reach of HIV-prevention services. An mHealth pilot intervention (titled "Despre Mine. Despre Noi." (DMDN) translated as "About Me. About Us."), which reduced Romanian GBM's risk for HIV infection while also reducing depression and alcohol abuse in an initial pre-post trial, is now ready for testing in a randomized controlled trial with a large national sample in the current study, entitled Comunică (translation: Communicate).

The Comunică intervention entails eight 60-minute live chat sessions delivered by trained counselors on a mobile study platform using motivational interviewing (MI) and cognitive-behavioral skills training (CBST). First, during pre-trial (months 1-5), in collaboration with a community advisory board consisting of GBM community members, GBM-affirmative physical and mental health providers, and a technical developer, the investigators will fine-tune the Comunică intervention based on the investigators' pilot findings and evaluation interviews, and expand the original DMDN education materials for an education attention condition (EAC) that will serve as control. Second, during the intervention phase (mos 6-45), the investigators will recruit, screen, assess, and randomize GBM at risk for HIV infection and alcohol abuse to either the Comunică intervention (n=163) or EAC (n=163). The conditions are content matched, and both are hosted on the study platform. While Comunică will consist of eight weekly mHealth live chat sessions, EAC will consist of eight self-administered educational modules. Third, during the follow-up phase (mos 8-55), the investigators will assess at 4, 8, and 12 months post-baseline, in a mobile fashion identical to the baseline, the primary outcome of condomless anal sex with male partners and secondary outcomes of alcohol abuse, depression, biologic HIV/STI infection, HIV/STI testing, and psychosocial mechanisms rooted in the Information-Motivation-Behavioral Skills (IMB) model (e.g., HIV/STI knowledge, condom use self-efficacy) and minority stress theory (e.g., identity concealment, internalized homophobia).

ELIGIBILITY:
Inclusion Criteria:

Gay and bisexual men (GMB) will be eligible if they report:

* Male sex at birth and current male identity;
* At least 16 years old;
* ≥ 1 act of condomless anal sex with an HIV-positive or status-unknown male partner in the prior month;
* ≥ 2 heavy drinking days in the prior month;
* Own a mobile device (smartphone, tablet, laptop); and
* Are confirmed to be HIV-negative upon testing at study baseline.

Exclusion Criteria:

* GMB will be excluded if they report past-year: a) psychiatric hospitalization; b) psychotic and manic symptoms; or c) current mood-stabilizing or anti-psychotic medication prescription
* Any condition that, in the principal investigators' judgment, interferes with safe study participation.

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Biological males at birth who currently identify as male
Enrollment: 300 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corina Lelutiu-Weinberger, PhD, Principal Investigator — Columbia University; John E. Pachankis, PhD, Principal Investigator — Yale University
Locations (1):
- Romanian Association against AIDS (ARAS), Bucharest, Ilfov, Romania

REFERENCES:
- [Derived] Lelutiu-Weinberger C, Filimon ML, Hoover D, Lixandru M, Hanu L, Dogaru B, Kovacs T, Fierbinteanu C, Ionescu F, Manu M, Maris A, Pana E, Dorobantescu C, Streinu-Cercel A, Pachankis JE. An mHealth Intervention for Gay and Bisexual Men's Mental, Behavioral, and Sexual Health in a High-Stigma, Low-Resource Context (Project Comunica): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 May 6;13:e52853. doi: 10.2196/52853. PMID 38709550
- [Derived] Lelutiu-Weinberger C, Filimon M, Hoover D, Lixandru M, Hanu L, Dogaru B, Kovaks T, Fierbinteanu C, Ionescu F, Manu M, Maris A, Pana E, Dorobantescu C, Streinu-Cercel A, Pachankis J. A randomized controlled trial of an mHealth intervention for gay and bisexual men's mental, behavioral, and sexual health in a high-stigma, low-resource context: Project Comunica protocol. Res Sq [Preprint]. 2023 Jun 26:rs.3.rs-3008174. doi: 10.21203/rs.3.rs-3008174/v1. PMID 37461458

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Comunică | Education Attention Control (EAC)
Started | 149 | 151
Completed | 149 | 151
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comunică | Education Attention Control (EAC) | Total
Number analyzed (Participants) | 149 | 151 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.93 (6.55) | 25.87 (7.38) | 25.40 (6.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 149 | 151 | 300
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Romanian | 137 | 137 | 274
  Hungarian | 10 | 10 | 20
  Roma | 1 | 2 | 3
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Romania | 149 | 151 | 300
Sexual orientation [Count of Participants; unit: Participants]
  Gay | 97 | 105 | 202
  Bisexual | 49 | 41 | 90
  Heterosexual | 0 | 0 | 0
  Queer | 1 | 1 | 2
  Pansexual | 1 | 1 | 2
  Asexual | 0 | 0 | 0
  Demisexual | 0 | 0 | 0
  Uncertain / don't know for sure | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-reported Condomless Anal Sex (CAS) Acts in the Last 30 Days
Description: Timeline Followback for Online Use (TLFB), which assesses sexual behavior (condomless anal sex acts) in the past month. It collects retrospective day-level data and has been validated for online self-administration.
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: Some participants were lost to follow-up, and in some cases participants did not provide data for certain outcomes on the self-administered surveys. Therefore, at some timepoints, "Number Analyzed" may be less that 149 for Comunica arm and 151 for Education Attention Control arm.
Measure: Mean (Standard Deviation); unit: condomless anal sex acts
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
condomless anal sex acts
  Baseline | 5.03 (5.47) | 6.40 (8.33)
  4 months: number analyzed (Participants) | 132 | 131
  4 months | 3.14 (7.01) | 2.37 (5.02)
  8 months: number analyzed (Participants) | 125 | 122
  8 months | 3.35 (6.58) | 2.60 (6.72)
  12 months: number analyzed (Participants) | 136 | 126
  12 months | 2.35 (4.65) | 3.15 (7.43)

2. Primary Outcome: Number of Self-reported Days With Heavy Alcohol Use in the Last 30 Days
Description: The Timeline Followback for Online Use (TLFB) tool will also ask participants to report occasions of heavy alcohol use (5 or more drinks) alone, and before/during sex, in the previous 30 days.
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days with heavy alcohol use
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
days with heavy alcohol use
  Baseline | 5.74 (4.98) | 5.32 (4.39)
  4 months: number analyzed (Participants) | 132 | 131
  4 months | 3.85 (3.84) | 3.06 (4.01)
  8 months: number analyzed (Participants) | 125 | 122
  8 months | 3.25 (3.81) | 2.80 (4.23)
  12 months: number analyzed (Participants) | 136 | 126
  12 months | 2.78 (3.68) | 2.48 (3.90)

3. Secondary Outcome: Score on Alcohol Use Disorders Identification Test (AUDIT-C)
Description: The Alcohol Use Disorders Identification Test (AUDIT-C) is a 3-item screening tool use to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Participants will report on standard drinks. The total score range is 0 to 12 (each item is scored 0-4), where an overall score of 4 or more is considered to indicate hazardous or harmful alcohol use. Higher scores indicate more hazardous/harmful alcohol use (i.e., a worse outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 5.14 (2.07) | 5.10 (2.03)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 4.24 (2.00) | 4.20 (2.14)
  8 months: number analyzed (Participants) | 131 | 125
  8 months | 4.05 (2.03) | 3.86 (1.99)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 3.94 (2.06) | 3.75 (1.88)

4. Secondary Outcome: Score on Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Center for Epidemiologic Studies Depression Scale (CES-D) is a self-report, standardized measure for depressive symptoms. It consists of 20 items in which respondents rate how frequently each item applied to them over the course of the past week. Ratings for each item are based on a 4-point Likert scale ranging from 0="rarely or none of the time (less than 1 day)" to 3="most or all of the time (5-7 days)". Item scores are summed to obtain an overall score from 0 to 60, where higher scores mean more depressive symptoms (i.e., a worse outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 22.06 (10.91) | 21.44 (13.83)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 17.30 (10.32) | 18.66 (11.96)
  8 months: number analyzed (Participants) | 131 | 125
  8 months | 17.80 (12.50) | 17.90 (12.25)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 16.82 (12.02) | 16.64 (11.83)

5. Secondary Outcome: Score on Beck's Anxiety Inventory (BAI)
Description: Beck's Anxiety Inventory (BAI) is a brief self-report measure of anxiety with a focus on somatic symptoms of anxiety that was developed as a measure adept at discriminating between anxiety and depression. It consists of 21 items and respondents indicate how much they have been bothered by each symptom over the past week. Responses to each item are rated on a 4-point Likert scale and range from 0="not at all" to 3="severely". Item scores are summed to obtain an overall score from 0 to 63, where higher scores indicate more anxiety symptoms (i.e., worse outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 15.20 (9.80) | 15.64 (10.04)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 10.73 (8.93) | 11.64 (9.69)
  8 months: number analyzed (Participants) | 131 | 125
  8 months | 9.55 (9.53) | 11.02 (10.51)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 9.98 (9.91) | 9.94 (9.98)

6. Other Pre Specified Outcome: Score on HIV Knowledge Questionnaire
Description: The HIV Knowledge Questionnaire is a 13-item, brief self-report measure of HIV-related knowledge. Respondents read each statement about HIV and indicate whether they think the statement is true or false, or they indicate that they "don't know." Responses are scored 0 (incorrect or unsure) or 1 (correct), and results are summed to obtain the number of statements correctly identified as true or false. The total score ranges from 0 to 13, where a higher score indicates more correct responses (i.e., better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 10.34 (1.96) | 10.50 (2.39)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 11.29 (1.57) | 11.83 (1.58)
  8 months: number analyzed (Participants) | 131 | 125
  8 months | 11.47 (1.87) | 11.78 (1.73)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 11.59 (1.51) | 12.06 (1.24)

7. Other Pre Specified Outcome: Score on Alcohol Effects Questionnaire
Description: Alcohol-related knowledge was measured through an 8-item version of a questionnaire featuring 8 true/false statements about alcohol (e.g., "A person cannot become an alcoholic by just drinking beer"). Responses were scored as either 0 (incorrect answer or "I don't know") or 1 (correct answer) and summed to obtain a final score from 0 to 8, where a higher score indicates a more correct responses (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 5.60 (1.40) | 5.60 (1.24)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 5.66 (1.45) | 6.05 (1.28)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 5.62 (1.58) | 5.94 (1.61)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 5.60 (1.63) | 6.37 (1.39)

8. Other Pre Specified Outcome: SOCRATES (Stages of Change Readiness and Treatment Eagerness Scale) - Problem Recognition Subscore
Description: The SOCRATES (Stages of Change Readiness and Treatment Eagerness Scale) is a 19-item, self-administered instrument designed to assess client motivation to change drinking-related behavior. It is made up of three subscales: Problem Recognition (score range 7 to 35), Ambivalence (score range is 4 to 20), and Taking Steps (score range is 8 to 40). Respondents rate their agreement with each item on a 5-point Likert-type scale (from 1=strongly disagree to 5=strongly agree), and items within each subscale are summed to obtain three subscores. A higher Problem Recognition subscore indicates a higher degree of recognition of one's problems related to their drinking (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 13.92 (6.38) | 13.93 (5.90)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 12.72 (6.31) | 12.68 (5.69)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 11.58 (5.77) | 12.07 (6.10)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 11.40 (6.17) | 11.55 (5.82)

9. Other Pre Specified Outcome: SOCRATES (Stages of Change Readiness and Treatment Eagerness Scale) - Ambivalence Subscore
Description: The SOCRATES (Stages of Change Readiness and Treatment Eagerness Scale) is a 19-item, self-administered instrument designed to assess client motivation to change drinking-related behavior. It is made up of three subscales: Problem Recognition (score range 7 to 35), Ambivalence (score range is 4 to 20), and Taking Steps (score range is 8 to 40). Respondents rate their agreement with each item on a 5-point Likert-type scale (from 1=strongly disagree to 5=strongly agree), and items within each subscale are summed to obtain three subscores. A higher Ambivalence subscore indicates a higher degree of ambivalence (e.g., openness to reflection) related to their drinking (as opposed to unawareness) (i.e., higher scores mean a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 8.85 (4.26) | 8.91 (4.05)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 7.88 (3.99) | 7.92 (4.01)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 7.02 (3.73) | 7.16 (3.91)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 6.94 (4.00) | 7.25 (3.94)

10. Other Pre Specified Outcome: SOCRATES (Stages of Change Readiness and Treatment Eagerness Scale) - Taking Steps Subscore
Description: The SOCRATES (Stages of Change Readiness and Treatment Eagerness Scale) is a 19-item, self-administered instrument designed to assess client motivation to change drinking-related behavior. It is made up of three subscales: Problem Recognition (score range 7 to 35), Ambivalence (score range is 4 to 20), and Taking Steps (score range is 8 to 40). Respondents rate their agreement with each item on a 5-point Likert-type scale (from 1=strongly disagree to 5=strongly agree), and items within each subscale are summed to obtain three subscores. A higher Taking Steps subscore indicates the individual is making attempts to change their drinking (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 16.74 (7.29) | 17.57 (6.90)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 17.96 (9.20) | 18.02 (8.27)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 16.09 (8.56) | 15.79 (7.84)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 16.51 (9.40) | 16.34 (8.63)

11. Other Pre Specified Outcome: Decisional Balance (Motivation to Use Condoms): Importance of Statements for Sex Without Condoms
Description: The Decisional Balance Scale assesses perceived benefits of sex with and without condoms. Responses to the 18-item scale assessed the benefits (e.g., "Sex without a condom is more spontaneous") and costs (e.g., "I feel guilty after having sex without a condom") of lack of condom use, yielding two subscales. Each participant was asked to rate how important each benefit and cost statement would be when deciding whether to use a condom for anal sex from 1="not at all important" to 5="extremely important"). Responses for each subscore ("Importance of statements for sex without condoms" and "Importance of statements against sex without condoms") are averaged to obtain two final subscores that range from 1 to 5. A higher "Importance of statements for sex without condoms" subscore indicates greater importance assigned to benefits of condomless anal sex (i.e., a worse outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 2.99 (0.77) | 3.00 (0.67)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 2.49 (0.82) | 2.69 (0.78)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 2.46 (0.87) | 2.61 (0.82)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 2.42 (0.85) | 2.59 (0.80)

12. Other Pre Specified Outcome: Decisional Balance (Motivation to Use Condoms): Importance of Statements Against Sex Without Condoms
Description: The Decisional Balance Scale assesses perceived benefits of sex with and without condoms. Responses to the 18-item scale assessed the benefits (e.g., "Sex without a condom is more spontaneous") and costs (e.g., "I feel guilty after having sex without a condom") of lack of condom use, yielding two subscales. Each participant was asked to rate how important each benefit and cost statement would be when deciding whether to use a condom for anal sex from 1="not at all important" to 5="extremely important"). Responses for each subscore ("Importance of statements for sex without condoms" and "Importance of statements against sex without condoms") are averaged to obtain two final subscores that range from 1 to 5. A higher "Importance of statements against sex without condoms" subscore indicates greater importance assigned to costs of condomless anal sex (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 3.20 (0.74) | 3.15 (0.81)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 3.26 (0.78) | 3.27 (0.75)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 3.23 (0.80) | 3.27 (0.80)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 3.16 (0.79) | 3.17 (0.79)

13. Other Pre Specified Outcome: Self-Efficacy for Safer Sex Questionnaire
Description: The Self-Efficacy for Safer Sex Questionnaire is a 13-item scale that measures behavioral self-efficacy skills to increase condom use. Response options for each item range from 1="not at all confident" to 5="extremely confident" in regards to participants' confidence in avoiding condomless sex and/or negotiating condom use. Item scores are summed to obtain an overall score from 1 to 65, where a higher score indicates greater confidence in avoiding condomless sex (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 37.38 (9.47) | 37.03 (10.80)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 44.95 (12.29) | 42.86 (12.55)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 45.13 (12.90) | 43.84 (12.10)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 46.01 (13.62) | 43.05 (12.62)

14. Other Pre Specified Outcome: Confidence in Reducing Alcohol Use (Drug-Taking Confidence Questionnaire) - Urges/Temptations To Use Subsore
Description: The Drug-Taking Confidence Questionnaire is a 50-item scale that measures behavioral self-efficacy skills to reduce alcohol use. An abbreviated 15-item version was used, which consists of the following three subscales from the original questionnaire: Urges/Temptations to Use (score range is 5 to 30), Social Pressure to Use (score range is 5 to 30), and Pleasant Times with Others (score range is 5 to 30). Responses to each item are rated from 1="not at all" to 6="completely", representing the level of confidence participants have in resisting alcohol use in each situation. Item scores within each subscale are summed to obtain the three subscores ranging from 5-30. A higher Urges/Temptations To Use subscore reflects greater confidence in resisting alcohol use when experiencing urges/temptations to use it (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 month post-baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 19.09 (7.39) | 18.50 (7.26)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 22.08 (6.68) | 20.64 (7.23)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 24.73 (6.29) | 25.74 (4.71)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 25.69 (5.43) | 25.48 (4.98)

15. Other Pre Specified Outcome: Confidence in Reducing Alcohol Use (Drug-Taking Confidence Questionnaire) - Social Pressure To Use Subscore
Description: The Drug-Taking Confidence Questionnaire is a 50-item scale that measures behavioral self-efficacy skills to reduce alcohol use. An abbreviated 15-item version was used, which consists of the following three subscales from the original questionnaire: Urges/Temptations to Use (score range is 5 to 30), Social Pressure to Use (score range is 5 to 30), and Pleasant Times with Others (score range is 5 to 30). Responses to each item are rated from 1="not at all" to 6="completely", representing the level of confidence participants have in resisting alcohol use in each situation. Item scores within each subscale are summed to obtain the three subscores ranging from 5-30. A higher Social Pressure to Use subscore reflects greater confidence in resisting alcohol use when under social pressure to use it (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8-months post-baseline, and 12 months post-baseline.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 16.13 (7.51) | 16.10 (7.24)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 18.83 (6.84) | 18.98 (7.67)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 23.17 (7.49) | 24.13 (6.42)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 23.83 (6.34) | 24.11 (5.96)

16. Other Pre Specified Outcome: Confidence in Reducing Alcohol Use (Drug-Taking Confidence Questionnaire) - Pleasant Times With Others Subscore
Description: The Drug-Taking Confidence Questionnaire is a 50-item scale that measures behavioral self-efficacy skills to reduce alcohol use. An abbreviated 15-item version was used, which consists of the following three subscales from the original questionnaire: Urges/Temptations to Use (score range is 5 to 30), Social Pressure to Use (score range is 5 to 30), and Pleasant Times with Others (score range is 5 to 30). Responses to each item are rated from 1="not at all" to 6="completely", representing the level of confidence participants have in resisting alcohol use in each situation. Item scores within each subscale are summed to obtain the three subscores ranging from 5-30. A higher Pleasant Times With Others subscore reflects greater confidence in resisting alcohol use in situations of experiencing pleasant times with others (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 16.31 (7.15) | 15.18 (7.03)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 17.92 (6.74) | 18.47 (7.76)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 23.19 (6.93) | 24.33 (5.67)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 23.67 (6.44) | 23.68 (6.22)

17. Other Pre Specified Outcome: Score on Gay-Related Rejection Sensitivity Scale
Description: The Gay-Related Rejection Sensitivity Scale is used to measure rejection sensitivity around one's sexuality. The scale consists of 14 interpersonal situations in which such rejection may be perceived (e.g., "You bring a male partner to a family reunion. Two of your old-fashioned aunts don't come talk to you even though they see you"), each followed by a question of anxiety (e.g., "How concerned or anxious would you be that they don't talk to you because of your sexual orientation?") and likelihood (e.g., "How likely is it that they didn't talk to you because of your sexual orientation?") of gay-related rejection occurring in this case, each scored from 1="very unconcerned/unlikely" to 6="very concerned/likely". The product of the likelihood and anxiety subscales for each of the 14 items were then averaged together to achieve an overall score. The overall score ranges from 1 to 36, where a higher score indicates greater gay-related rejection sensitivity (i.e., a worse outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 13.44 (7.30) | 13.64 (7.58)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 10.58 (6.94) | 11.44 (7.88)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 9.57 (7.65) | 9.83 (7.40)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 8.81 (7.44) | 8.92 (7.57)

18. Other Pre Specified Outcome: Score on Rathus Assertiveness Schedule
Description: The Rathus Assertiveness Schedule is a 30-item self-report which measure assertive behaviors. The items include statements like "Most people seem to be more aggressive and assertive than I am", "When I am asked to do something, I insist upon knowing why" etc. The responses ranges from -3="very uncharacteristic of me" to 3="very characteristic of me". Items 1, 2, 4, 5, 9, 11-17, 19, 23, 24, 26, and 30 are reverse-coded and the resulting 30 items are summed to attain a continuous score from -90 to 90, where a higher score indicates greater assertiveness (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline: number analyzed (Participants) | 148 | 150
  Baseline | 6.71 (24.38) | 7.57 (24.25)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 11.49 (24.19) | 9.45 (24.03)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 11.02 (22.85) | 10.05 (25.84)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 10.93 (23.17) | 11.79 (24.98)

19. Other Pre Specified Outcome: Lesbian, Gay, and Bisexual Identity Scale (LGBIS) - Concealment Motivation Subscore
Description: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) is a 27-item, self-reported measure that assesses an individual's sexual minority identity across eight dimensions/subscales: acceptance concerns, concealment motivation, identity uncertainty, internalized homonegativity, difficulty with the identity development process, identity superiority, identity affirmation, and identity centrality. Responses to items were scored from 1="disagree strongly" to 6="agree strongly", with items 11 and 23 being reverse-coded. Items within each subscale averaged to obtain eight final subscores. The concealment motivation subscore ranges from 1-6 with higher scores indicating a greater degree of motivation to conceal one's sexual minority identity.
Time Frame: Measured at baseline, 4 months post-intervention, 8 months post-intervention, and 12 months post-intervention.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 4.36 (1.22) | 4.36 (1.29)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 4.25 (1.28) | 4.22 (1.21)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 4.19 (1.24) | 4.29 (1.34)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 4.23 (1.28) | 4.17 (1.27)

20. Other Pre Specified Outcome: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) - Internalized Homonegativity Subscore
Description: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) is a 27-item, self-reported measure that assesses an individual's sexual minority identity across eight dimensions/subscales: acceptance concerns, concealment motivation, identity uncertainty, internalized homonegativity, difficulty with the identity development process, identity superiority, identity affirmation, and identity centrality. Responses to items were scored from 1="disagree strongly" to 6="agree strongly", with items 11 and 23 being reverse-coded. Items within each subscale averaged to obtain eight final subscores. The internalized homonegative subscore ranges from 1-6 with higher scores indicating greater internalized homonegativity (i.e., a worse outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 2.40 (1.30) | 2.26 (1.24)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 2.26 (1.22) | 2.18 (1.22)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 2.34 (1.41) | 2.20 (1.32)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 2.25 (1.27) | 2.19 (1.28)

21. Other Pre Specified Outcome: Lesbian, Gay, and Bisexual Identity Scale (LGBIS) - Acceptance Concerns Subscore
Description: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) is a 27-item, self-reported measure that assesses an individual's sexual minority identity across eight dimensions/subscales: acceptance concerns, concealment motivation, identity uncertainty, internalized homonegativity, difficulty with the identity development process, identity superiority, identity affirmation, and identity centrality. Responses to items were scored from 1="disagree strongly" to 6="agree strongly", with items 11 and 23 being reverse-coded. Items within each subscale averaged to obtain eight final subscores. The acceptance concerns subscore ranges from 1-6 with higher scores indicating more acceptance concerns (i.e., a worse outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 3.69 (1.30) | 3.47 (1.25)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 3.46 (1.21) | 3.26 (1.35)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 3.35 (1.27) | 3.20 (1.38)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 3.31 (1.31) | 3.02 (1.26)

22. Other Pre Specified Outcome: Lesbian, Gay, and Bisexual Identity Scale (LGBIS) - Identity Uncertainty Subscore
Description: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) is a 27-item, self-reported measure that assesses an individual's sexual minority identity across eight dimensions/subscales: acceptance concerns, concealment motivation, identity uncertainty, internalized homonegativity, difficulty with the identity development process, identity superiority, identity affirmation, and identity centrality. Responses to items were scored from 1="disagree strongly" to 6="agree strongly", with items 11 and 23 being reverse-coded. Items within each subscale averaged to obtain eight final subscores. The identity uncertainty subscore ranges from 1-6 with higher scores indicating a greater degree of uncertainty about one's sexual minority identity.
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 2.09 (1.13) | 2.05 (1.19)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 2.01 (1.15) | 2.09 (1.21)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 1.93 (1.15) | 2.06 (1.25)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 1.90 (1.08) | 1.93 (1.20)

23. Other Pre Specified Outcome: Lesbian, Gay, and Bisexual Identity Scale (LGBIS) - Difficult Process Subscore
Description: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) is a 27-item, self-reported measure that assesses an individual's sexual minority identity across eight dimensions/subscales: acceptance concerns, concealment motivation, identity uncertainty, internalized homonegativity, difficulty with the identity development process, identity superiority, identity affirmation, and identity centrality. Responses to items were scored from 1="disagree strongly" to 6="agree strongly", with items 11 and 23 being reverse-coded. Items within each subscale averaged to obtain eight final subscores. The difficult process subscore ranges from 1-6 with higher scores indicating the participant has been having a more difficult time accepting their sexual minority identity.
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 3.66 (1.40) | 3.42 (1.41)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 3.39 (1.34) | 3.31 (1.38)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 3.45 (1.35) | 3.29 (1.39)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 3.49 (1.36) | 3.24 (1.28)

24. Other Pre Specified Outcome: Lesbian, Gay, and Bisexual Identity Scale (LGBIS) - Identity Superiority Subscore
Description: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) is a 27-item, self-reported measure that assesses an individual's sexual minority identity across eight dimensions/subscales: acceptance concerns, concealment motivation, identity uncertainty, internalized homonegativity, difficulty with the identity development process, identity superiority, identity affirmation, and identity centrality. Responses to items were scored from 1="disagree strongly" to 6="agree strongly", with items 11 and 23 being reverse-coded. Items within each subscale averaged to obtain eight final subscores. The identity superiority subscore ranges from 1-6 with higher scores indicating the participant views people with a sexual minority identity as superior to heterosexual people.
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 2.21 (1.05) | 2.32 (1.03)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 2.18 (1.12) | 2.33 (1.07)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 2.24 (1.14) | 2.31 (1.11)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 2.23 (1.12) | 2.37 (1.19)

25. Other Pre Specified Outcome: Lesbian, Gay, and Bisexual Identity Scale (LGBIS) - Identity Affirmation Subscore
Description: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) is a 27-item, self-reported measure that assesses an individual's sexual minority identity across eight dimensions/subscales: acceptance concerns, concealment motivation, identity uncertainty, internalized homonegativity, difficulty with the identity development process, identity superiority, identity affirmation, and identity centrality. Responses to items were scored from 1="disagree strongly" to 6="agree strongly", with items 11 and 23 being reverse-coded. Items within each subscale averaged to obtain eight final subscores. The identity affirmation subscore ranges from 1-6 with higher scores indicating greater pride in one's sexual minority identity (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 4.27 (1.30) | 4.32 (1.21)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 4.31 (1.30) | 4.30 (1.24)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 4.13 (1.39) | 4.46 (1.26)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 4.21 (1.41) | 4.37 (1.36)

26. Other Pre Specified Outcome: Lesbian, Gay, and Bisexual Identity Scale (LGBIS) - Identity Centrality Subscore
Description: The Lesbian, Gay, and Bisexual Identity Scale (LGBIS) is a 27-item, self-reported measure that assesses an individual's sexual minority identity across eight dimensions/subscales: acceptance concerns, concealment motivation, identity uncertainty, internalized homonegativity, difficulty with the identity development process, identity superiority, identity affirmation, and identity centrality. Responses to items were scored from 1="disagree strongly" to 6="agree strongly", with items 11 and 23 being reverse-coded. Items within each subscale averaged to obtain eight final subscores. The identity centrality subscore ranges from 1-6 with higher scores indicating that one's sexual orientation is more central to one's personal identity.
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 3.65 (1.02) | 3.79 (1.18)
  4 months: number analyzed (Participants) | 134 | 132
  4 months | 3.63 (1.05) | 3.76 (1.16)
  8 months: number analyzed (Participants) | 130 | 125
  8 months | 3.62 (1.16) | 3.83 (1.17)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 3.61 (1.18) | 3.88 (1.18)

27. Other Pre Specified Outcome: Score on LGBT Victimization Scale
Description: The 10-item version of the LGBT Victimization Scale measures that assesses the frequency of experiences of victimization in the previous 3 months "because you are, or were thought to be, gay, lesbian, bisexual, or transgender." Items address verbal threats and insults, being chased, having property damaged, and being physically or sexually assaulted. Responses to each item/situation are scored from 0="never" to 3="3 or more times" and summed to obtain an overall score, which ranges from 0 to 30, where a higher score indicates higher frequency of victimization experiences (i.e., a worse outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 2.13 (3.24) | 2.30 (4.50)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 1.43 (3.25) | 1.57 (3.35)
  8 months: number analyzed (Participants) | 130 | 124
  8 months | 1.08 (3.23) | 1.37 (4.42)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 0.86 (2.40) | 0.87 (2.53)

28. Other Pre Specified Outcome: Score on Multidimensional Scale of Perceived Social Support (MSPSS)
Description: The Multidimensional Scale of Perceived Social Support (MSPSS) is a 12-item self-reported questionnaire designed to measure perceived social support from three sources: family, friends, and a significant other. Responses are scored from 1="very strongly disagree" to 7="very strongly agree" and averaged to obtain a final score that ranges from 1 to 7, where a higher score indicates higher perceived social support (i.e., a better outcome).
Time Frame: Measured at baseline, 4 months post-baseline, 8 months post-baseline, and 12 months post-baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comunică | Education Attention Control (EAC)
Number analyzed (Participants) | 149 | 151
score on a scale
  Baseline | 4.98 (1.27) | 4.81 (1.35)
  4 months: number analyzed (Participants) | 135 | 132
  4 months | 5.21 (1.16) | 4.95 (1.42)
  8 months: number analyzed (Participants) | 130 | 124
  8 months | 4.94 (1.43) | 5.01 (1.50)
  12 months: number analyzed (Participants) | 138 | 129
  12 months | 5.03 (1.40) | 5.10 (1.50)

ADVERSE EVENTS:
Time Frame: During an assessment or counseling session, from baseline survey to 12-months post randomization
Description: Participants were assessed as soon as a trigger was sent to the team by a score in a survey, or an event was discovered during a counseling session.
Arm/Group | Comunică | Education Attention Control (EAC)
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/151
Serious Adverse Events (participants affected / at risk) | 2/149 | 0/151
Other Adverse Events (participants affected / at risk) | 14/149 | 16/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Comunică (N=149) | Education Attention Control (EAC) (N=151)
Suicide attempt (Psychiatric disorders) | 2 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Comunică (N=149) | Education Attention Control (EAC) (N=151)
Suicidal ideation (Psychiatric disorders) | 14 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-02-15): https://cdn.clinicaltrials.gov/large-docs/53/NCT03912753/Prot_001.pdf
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/53/NCT03912753/SAP_000.pdf